CLINICAL TRIAL: NCT03606460
Title: A Phase IIIb, Open-Label Study To Evaluate The Safety And Tolerability Of Shorter Infusions Of Ocrelizumab In Patients With Primary Progressive And Relapsing Multiple Sclerosis
Brief Title: A Study to Evaluate the Safety of Administering Ocrelizumab Per a Shorter Infusion Protocol in Participants With Primary Progressive Multiple Sclerosis (PPMS) and Relapsing Multiple Sclerosis (RMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40638
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): This cohort will examine the effect of administering ocrelizumab per a shorter infusion protocol for Dose 2 or Dose 3. Participants who have already received one or two doses of ocrelizumab according to the approved infusion protocol and have reported no serious infusion-related reactions (IRRs) will be enrolled. They will then receive the next infusion of ocrelizumab (Dose 2 or Dose 3) at a dosage of 600 milligram (mg) over the course of approximately 2 hours. Dose 2 is administered at Week 24, Dose 3 is administered at Week 48 after initial infusion.
  Interventions: Drug: Ocrelizumab Dose 2 and Dose 3
- Cohort 2 (Experimental): This cohort will examine the effect of administering ocrelizumab per a shorter infusion protocol for the second infusion of Dose 1. Ocrelizumab-naïve participants will be enrolled who, after receiving Dose 1 of ocrelizumab at the approved rate have no reported serious IRRs, will then receive the second 300-mg shorter infusion over approximately 1.5 hours.
  Interventions: Drug: Ocrelizumab Dose 1

INTERVENTIONS:
Drug: Ocrelizumab Dose 1 — 300 mg infusion administered to ocrelizumab-naive participants per approved protocol (over approximately 2.5 hours or longer) as per standard of care followed by a second 300 mg shorter infusion over approximately 1.5 hours.
  Arms: Cohort 2
Drug: Ocrelizumab Dose 2 and Dose 3 — 600 mg infusion of ocrelizumab administered at a shorter rate (i.e. over the course of approximately 2 hours) at Week 24 and at Week 48
  Arms: Cohort 1

SUMMARY:
This study is an open-label, non-randomized study to evaluate rate and severity of infusion-related reactions (IRRs) of ocrelizumab infused over a shorter time period than the approved administration rate in participants with PPMS or RMS in the United States (U.S.). Participants will be enrolled into two cohorts. Cohort 1 will examine the effect of administering ocrelizumab per a shorter infusion protocol for Dose 2 or Dose 3. This cohort will consist of patients who have already received one or two doses of ocrelizumab according to the approved infusion protocol (i.e., per the currently U.S. label) and have reported no serious IRRs and who will then receive the next infusion of ocrelizumab at a higher rate in order to deliver 600 mg over the course of approximately 2 hours. Cohort 2 will examine the effect of administering ocrelizumab per a shorter infusion protocol for the second infusion of Dose 1. This cohort will consist of ocrelizumab naïve patients who, after receiving Infusion 1/Dose 1 of ocrelizumab at the approved rate (300 mg over approximately 2.5 hours or longer) have no reported serious IRRs, will then receive the second 300-mg shorter infusion over approximately 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive ocrelizumab per the United States Package Insert (USPI)
* Able to comply with the study protocol, in the investigator's judgment
* Age 18-55 years, inclusive
* Have a diagnosis of PPMS or RMS, confirmed per the revised 2017 McDonald criteria
* Expanded Disability Status Scale (EDSS) score of 0 to 6.5, inclusive
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last dose of study treatment (per the USPI)

Exclusion Criteria:

* Experienced serious IRR(s)
* History of life-threatening infusion reaction to ocrelizumab
* Known presence of other neurological disorders
* Pregnancy or lactation, or intention to become pregnant during the study
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Significant, uncontrolled disease, such as cardiovascular (including cardiac arrhythmia), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine, and gastrointestinal or any other significant disease that may preclude patient from participating in the study
* Congestive heart failure
* Known active bacterial, viral, fungal, mycobacterial infection or other infection or any severe episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit
* History of or currently active primary or secondary immunodeficiency
* History or known presence of recurrent or chronic infection (e.g., HIV, syphilis, tuberculosis)
* History of recurrent aspiration pneumonia requiring antibiotic therapy
* History of malignancy, including solid tumors and hematological malignancies,except basal cell, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix of the uterus that have been excised with clear margins
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of alcohol or drug abuse within 24 weeks prior to enrollment
* Receipt of a live vaccine within 6 weeks prior to enrollment
* Systemic corticosteroid therapy within 4 weeks prior to enrollment
* Contraindications to or intolerance of oral or IV corticosteroids, including IV methylprednisolone (or equivalent steroid) administered according to the country label
* Treatment with alemtuzumab
* Treatment with a B-cell targeted therapies other than ocrelizumab
* Treatment with a drug that is experimental
* Abnormal laboratory results per local laboratory standards and investigator assessment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - University of Colorado; Anschutz Medical Campus Department of Neurology, Aurora, Colorado
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - Cleveland Clinic Fndn, Cleveland, Ohio
  - Ohio Health Research Institute Grant Medical Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation; MS Center of Excellence, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Vollmer TL, Cohen JA, Alvarez E, Nair KV, Boster A, Katz J, Pardo G, Pei J, Raut P, Merchant S, MacLean E, Pradhan A, Moss B. Safety results of administering ocrelizumab per a shorter infusion protocol in patients with primary progressive and relapsing multiple sclerosis. Mult Scler Relat Disord. 2020 Nov;46:102454. doi: 10.1016/j.msard.2020.102454. Epub 2020 Aug 18. PMID 33045496

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: This cohort examined the effect of administering ocrelizumab per a shorter infusion protocol for Dose 2 or Dose 3. Participants who had already received one or two doses of ocrelizumab according to the approved infusion protocol and had reported no serious infusion-related reactions (IRRs) were enrolled. They then received the next infusion of ocrelizumab (Dose 2 or Dose 3) at a dosage of 600 milligram (mg) over the course of approximately 2 hours. Dose 2 was administered at Week 24, Dose 3 was administered at Week 48 after initial infusion.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 95 | 46
Completed | 94 | 38
Not Completed | 1 | 8
Not completed — Lost to Follow-up | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 95 | 46 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.75 (8.80) | 41.07 (8.74) | 41.52 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 34 | 93
  Male | 36 | 12 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 88 | 41 | 129
  Unknown | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 8 | 16
  White | 86 | 35 | 121
  Multiple | 1 | 0 | 1
  Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Infusion-related Reaction (IRR) Treated With 600 mg IV Ocrelizumab
Description: This outcome measure evaluates the occurrence of severe infusion-related reaction (IRR) with ocrelizumab 600 mg intravenously (IV) administered over the course of 2 hours. Rate and frequency of NCI CTCAE v4.0 Grade 3 and 4 IRRs
Time Frame: During or within 24 hours of administration
Population: The Safety population was the same as the ITT population in this study. All enrolled participants received study treatment, hence treatment group comparability is not applicable. The analysis was conducted in Cohort 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 95
Percentage of Participants | 0 [0.0 to 3.8]

2. Secondary Outcome: Percentage of Participants With IRRs
Description: This outcome measure evaluates the occurrence of overall IRRs with ocrelizumab either 300mg or 600mg IV infusion. Rate and frequency of NCI CTCAE v4.0 Grade 1-4 IRRs.
Time Frame: During or within 24 hours of administration
Population: The Safety Population was defined as all enrolled participants who received any dose of study treatment, even if the infusion was incomplete. All enrolled participants received study treatment. The Safety population was the same as the ITT population in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 95 | 46
Percentage of Participants | 48.4 [38.0 to 58.9] | 10.9 [3.6 to 23.6]

3. Secondary Outcome: Percentage of Participants With IRRs Treated With the 300 mg Shorter Dose of Ocrelizumab
Description: This outcome measure evaluate the occurrence of severe IRRs with ocrelizumab 300 mg administered over the course of 1.5 hours. Rate and frequency of NCI CTCAE v4.0 Grade 3-4 IRRs.
Time Frame: During or within 24 hours of administration
Population: The Safety population was the same as the ITT population in this study. All enrolled participants received study treatment, hence treatment group comparability is not applicable. The analysis was conducted in Cohort 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 46
Percentage of Participants | 0 [0.0 to 7.7]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The Safety Population was defined as all enrolled participants who received any dose of study treatment, even if the infusion was incomplete. All enrolled participants received study treatment. The Safety population was the same as the ITT population in this study.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/46
Other Adverse Events (participants affected / at risk) | 46/95 | 7/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=95) | Cohort 2 (N=46)
Fatigue (General disorders) | 1 (1) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 46 (65) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03606460/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03606460/SAP_001.pdf